CLINICAL TRIAL: NCT04284345
Title: Diagnostic Accuracy of the Saline-induced Distal to Aortic Coronary Pressure Ratio Compared With Clinically Available Resting and Hyperemic Indices of Coronary Artery Stenosis Severity
Brief Title: Saline-induced Distal to Aortic Coronary Pressure Ratio vs. Resting and Hyperemic Indices of Coronary Artery Stenosis Severity
Acronym: SALINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, IGLESIAS Juan Fernando, Principal investigator, University Hospital, Geneva
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-00910
Record Dates: First submitted 2020-01-09; First posted 2020-02-25 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Coronary Stenosis
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Saline Pd/Pa (Experimental): Eligible subjects will undergo invasive coronary physiology measurements including whole cycle resting Pd/Pa, iFR, RFR, cFFR, Saline Pd/Pa and FFR
  Interventions: Procedure: Saline Pd/Pa

INTERVENTIONS:
Procedure: Saline Pd/Pa — Use of a ≥6F guiding catheter and the Verrata pressure guidewire. Administration of intracoronary nitroglycerin.
  Verrata normalisation and placement of the Verrata sensor ≥3 vessel-diameter beyond the stenosis.
  Whole cycle resting Pd/Pa and resting iFR measurements.
  Measurement of contrast FFR: record 5 baseline heart beats, injection of contrast media, 10 ml in the left coronary system, 8 ml in the right coronary system, measure minimal Pd/Pa under stable hyperaemia.
  Adenosine FFR: measurement: record 5 baseline heart beats, injection of intracoronary adenosine, 200 mcg in the left coronary system, 100 mcg in the right coronary system, measure minimal Pd/Pa under stable hyperaemia.
  Saline-induced Pd/Pa measurement: record 5 baseline heart beats, injection of saline using the ACIST system during 5 heart beats, measure minimal Pd/Pa under stable hyperaemia.
  Perform pressure guidewire pullback and check for drift: drift ±0.02 is accepted, if ≥0.03, repeat measurement.

SUMMARY:
The presence of inducible myocardial ischemia is considered as the prerequisite for the clinical benefit of coronary revascularization. In this regard, the introduction of invasive pressure-derived physiological indices to guide myocardial revascularization represented a major breakthrough for the treatment of patients with coronary artery disease (CAD), by moving the focus of coronary revascularization from anatomy to physiology . The main premise of coronary physiology is to permit determination of the functional significance of individual stenoses on a per-vessel basis, measurable at the time of clinical decision-making process, thus providing an objective marker to identify ischemic lesions, and therefore patients, most likely to benefit from coronary revascularization .

Fractional flow reserve (FFR) is the most widely used pressure-derived invasive physiological index for coronary lesion assessment in contemporary clinical practice. FFR is calculated as the ratio of the mean distal coronary pressure (Pd) to the mean proximal coronary pressure (Pa) across a stenosis during maximal hyperaemia, a condition that is commonly achieved by the intracoronary or intravenous administration of a potent vasodilator agent, such as adenosine. Based on the results of landmark clinical trials, most recent guidelines recommend the use of FFR to identify hemodynamically significant coronary lesions in patients with stable CAD. Despite this, the worldwide adoption of FFR into current clinical practice remains limited , accounting for only 9.8% of coronary procedures in Switzerland . Potential reasons for the low adoption rate of coronary physiology include technical challenges and time consumption related to FFR measurements, inadequate or lack of reimbursement, physician preferences, patient-related discomfort, contraindications and costs associated with adenosine, or in certain countries, no availability of adenosine.

The low use of FFR in clinical practice provided a rationale for the development of new invasive physiology indices. By negating the need for administration of pharmacologic agents such as adenosine, saving time, and reducing costs and side effects, hyperaemia-free pressure-derived physiological indices were developed to increase adoption of physiology-guided coronary revascularization into routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥18 years of age.
* Subject must be willing to sign a Patient Informed Consent (PIC).
* Coronary artery disease with over 50% angiographic diameter stenosis on visual assessment, undergoing clinically indicated invasive physiological assessment by means of FFR.
* Assessment of non culprit arteries with over 50% angiographic diameter stenosis on visual assessment, in patients presenting with NSTEMI.

Exclusion Criteria:

* Pregnant and/or breastfeeding females.
* Known allergies to: heparin, contrast medium, adenosine.
* Contra-indication to adenosine.
* Severe renal failure (eGFR ≤ 30 ml/min/m2).
* Ostial stenosis in both the left and right coronary arteries.
* Presence of a chronic total occlusion.
* History of coronary artery bypass graft.
* Acute coronary syndrome.
* Acute myocardial infarction within the preceding two weeks.
* Severe valvular heart disease.
* Left main disease.
* Documented left ventricular ejection fraction (LVEF) ≤30% as documented within maximum 6 months prior to the procedure.
* Decompensated congestive heart failure.
* Extreme hypotension (systolic blood pressure <100 mmHg)
* Extreme bradycardia (<40 bpm).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Saline Pd/Pa ratio | during the coronarography procedure
  As the patient will undergo invasive physiological assessment of an angiographic intermediate stenosis with fractional flow reserve (FFR), as per ESC guidelines recommendation (class of recommendation I, level of evidence A), we will perform measurement of saline Pd/Pa with the same pressure guidewire, requiring an additional 3-5 minutes and injection of 10 ml of saline.
Contrast Fractional Flow Reserve (FFR) | during the coronarography procedure
  As the patient will undergo invasive physiological assessment of an angiographic intermediate stenosis with fractional flow reserve (FFR), as per ESC guidelines recommendation (class of recommendation I, level of evidence A), we will perform measurement of contrast fractional flow reserve (FFR) with the same pressure guidewire, requiring an additional 3-5 minutes and injection of 10 ml of contrast.
Adenosine Fractional Flow Reserve (FFR) | during the coronarography procedure
  The patient will undergo invasive physiological assessment of an angiographic intermediate stenosis with fractional flow reserve (FFR), as per ESC guidelines recommendation (class of recommendation I, level of evidence A).
Resting Pd/Pa ratio | during the coronarography procedure
  As the patient will undergo invasive physiological assessment of an angiographic intermediate stenosis with fractional flow reserve (FFR), as per ESC guidelines recommendation (class of recommendation I, level of evidence A), we will perform measurement of Pd/Pa with the same pressure guidewire, requiring an additional 3-5 minutes.
Instantaneous wave-free ratio (iFR) | during the coronarography procedure
  The patient will undergo invasive physiological assessment of an angiographic intermediate stenosis with instantaneous wave-free ratio (iFR), as per ESC guidelines recommendation (class of recommendation I, level of evidence A).

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland